CLINICAL TRIAL: NCT04225247
Title: Efficacy of Seventh Generation Bonding Agents as Short-Term Desensitizers Among Patients With Hypersensitivity A Randomized Clinical Trial
Brief Title: Efficacy of Seventh Generation Bonding Agents as Short-Term Desensitizers Among Patients With Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sumaiya Shabbir, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2358847
Record Dates: First submitted 2019-12-27; First posted 2020-01-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin hypersensitivity; Gingival Recession; Bonding Agents
MeSH Terms: conditions — Dentin Sensitivity; Gingival Recession | interventions — Bifluorid 12; Xeno V

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group-I Single Bond Universal (Active Comparator): it is a seventh generation bonding agent used as desensitizer, manufactured by 3M ESPE.
  applied on the affected surface of the group-I participants.
  Interventions: Drug: Single Bond Universal
- Group-II Xeno V+ (Active Comparator): it is a seventh generation bonding agent used as desensitizer, manufactured by Dentsply.
  applied on the affected surface of the group-II participants.
  Interventions: Drug: Xeno V+
- Group-III Bifluorid 12 (Placebo Comparator): it is a fluoride varnish used as desensitizer, manufactured by VOCO. applied on the affected surface of the group-III participants.
  Interventions: Drug: Bifluorid 12

INTERVENTIONS:
Drug: Single Bond Universal — Single bond universal (by 3M ESPE) is a seventh generation bonding agents used as desensitizers in the present study.
  Arms: Group-I Single Bond Universal
Drug: Bifluorid 12 — it is a fluoride varnish by VOCO.
  Arms: Group-III Bifluorid 12
Drug: Xeno V+ — Xeno V+ (by Dentsply) is a seventh generation bonding agents used as desensitizers in the present study.
  Arms: Group-II Xeno V+

SUMMARY:
The world lacks a gold standard treatment for treating dentin hypersensitivity. Fluoride varnish is most commonly used as a treatment but it causes temporary discoloration of tooth structure and may cause irritation or burning of gums when it comes in contact with gums. Seventh generation bonding agents are less technique sensitive and are easy to use. The present study aims to find out the better seventh generation bonding agent as a treatment option for sensitivity.

A total of 105 patients with dentin hypersensitivity are randomized into three groups. Scaling and root debridement are performed for all the groups. This study compares two seventh generation bonding agents and taking fluoride varnish as control group.

DETAILED DESCRIPTION:
Dentin hypersensitivity is a painful condition resulting from external stimulation of exposed vital dentin. Dentin gets exposed to the oral environment by multiple factors like gingival recession, erosion, attrition, abrasion, fractures, caries, and many more. The intra-tubular fluid movement of exposed tubules is believed to be the mechanism of hypersensitivity. Dentin bonding agents acts by occluding patent tubules, thus reducing hypersensitivity. Seventh generation combines etchant, primer and bonding agent into one solution and makes it easy to use.

After diagnosis of dentin hypersensitivity, the patients signed a consent form stating their voluntary participation in the research. The discomfort internal scale score and Schiff cold air sensitivity scale scores are recorded at baseline, immediately after the intervention, after 01 week and after 01 month. Discomfort internal scale score are recorded for every participant using dental explorer in the mesial and distal direction on the exposed surface of the affected teeth for tactile stimulation. For schiff cold air sensitivity scale scores an air syringe system was used to check the evaporative response on the affected teeth of the participants and the scores are recorded.

All the patients received scaling and root debridement as a standard protocol treatment. Dentin bonding agents and fluoride varnish are applied to the participants. All the participants are instructed to fast for two hours after the treatment. All the records are made on subjective response of patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of 18 to 45 years of age
* Hypersensitive teeth to air and tactile stimultaion
* Gingival recession of Miller Class I and II
* Score 1 of Silness and Loe Plaque index
* Participants who have no sysytemic illness
* Patients who agree to give consent were included in the study.

Exclusion Criteria:

* Carious teeth
* Fractured restoration or cracked teeth
* Teeth undergoing orthodontic or periodontal treatment at sensitive site
* Patients who had dental bleaching in last 03 months
* Patients taking pain killers
* Smokers
* Pregnant and nursing females were excluded from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-10-07 (Actual); Study Completion 2018-10-07 (Actual)

PRIMARY OUTCOMES:
Discomfort Internal Scale score | 1 month
  0 - No Pain
  1. - Mild
  2. - Moderate
  3. - Severe
  4. - Intolerable Pain
Schiff Cold Air Sensitivity Scale Score | 1 month
  Grade 0 - Subject does not respond to air stimulus. Grade 1 - Subject responds to air stimulus does not request discontinuation of stimulus.
  Grade 2- Subject responds to air stimulus and requests discontinuation or moves away from stimulus.
  Grade 3 - Subject responds to air stimulus, considers stimulus to be painful and requests discontinuation of stimulus.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu X, Liang B, Jin X, Fu B, Hannig M. Comparative in vivo study on the desensitizing efficacy of dentin desensitizers and one-bottle self-etching adhesives. Oper Dent. 2010 May-Jun;35(3):279-86. doi: 10.2341/09-346-C. PMID 20533627
- [Background] Ferrari M, Cagidiaco MC, Kugel G, Davidson CL. Clinical evaluation of a one-bottle bonding system for desensitizing exposed roots. Am J Dent. 1999 Oct;12(5):243-9. PMID 10649916
- [Background] Torres CR, Silva TM, Fonseca BM, Sales AL, Holleben P, Di Nicolo R, Borges AB. The effect of three desensitizing agents on dentin hypersensitivity: a randomized, split-mouth clinical trial. Oper Dent. 2014 Sep-Oct;39(5):E186-94. doi: 10.2341/13-057. Epub 2014 Apr 10. PMID 24720265
- [Background] Hajizadeh H, Nemati-Karimooy A, Majidinia S, Moeintaghavi A, Ghavamnasiri M. Comparing the effect of a desensitizing material and a self-etch adhesive on dentin sensitivity after periodontal surgery: a randomized clinical trial. Restor Dent Endod. 2017 Aug;42(3):168-175. doi: 10.5395/rde.2017.42.3.168. Epub 2017 Jul 21. PMID 28808633
- [Background] Panduric V, Knezevic A, Tarle Z, Sutalo J. The efficiency of dentine adhesives in treating non-caries cervical lesions. J Oral Rehabil. 2001 Dec;28(12):1168-74. doi: 10.1046/j.1365-2842.2001.00779.x. PMID 11874519
- [Background] Bartold PM. Dentinal hypersensitivity: a review. Aust Dent J. 2006 Sep;51(3):212-8; quiz 276. PMID 17037886
- [Background] Polderman RN, Frencken JE. Comparison between effectiveness of a low-viscosity glass ionomer and a resin-based glutaraldehyde containing primer in treating dentine hypersensitivity--a 25.2-month evaluation. J Dent. 2007 Feb;35(2):144-9. doi: 10.1016/j.jdent.2006.06.005. Epub 2006 Sep 14. PMID 16973252
- [Background] Schiff T, Dotson M, Cohen S, De Vizio W, McCool J, Volpe A. Efficacy of a dentifrice containing potassium nitrate, soluble pyrophosphate, PVM/MA copolymer, and sodium fluoride on dentinal hypersensitivity: a twelve-week clinical study. J Clin Dent. 1994;5 Spec No:87-92. PMID 8534380
- [Derived] Shabbir S, Ahmed S, Zaidi SJA, Riaz S, Sarwar H, Taqi M, Rahman Khan ZU. Efficacy of seventh generation bonding agents as desensitizers in patients with dentin hypersensitivity: a randomized clinical trial. BMC Oral Health. 2024 May 14;24(1):562. doi: 10.1186/s12903-024-04352-0. PMID 38745306